CLINICAL TRIAL: NCT02532361
Title: A Retrospective Analysis to Describe the Proportion of Hysterectomy After Female Sterilization With Hysteroscopic Device or Tubal Ligation Using Intermountain Healthcare Database in the US
Brief Title: Proportion of Hysterectomy After Female Sterilization
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18473
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Hysterectomy
Keywords: Sterilization; Hysteroscopic Device Placement; Tubal Ligation
MeSH Terms: interventions — Sterilization, Tubal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1 / Hysteroscopic device placement: Patients that had undergone sterilization through hysteroscopic device placement
  Interventions: Device: Hysteroscopic device placement including Essure (ESS305, BAY1454032)
- Cohort 2 / Tubal ligation: Patients that had undergone sterilization through tubal ligation
  Interventions: Procedure: Tubal ligation

INTERVENTIONS:
Device: Hysteroscopic device placement including Essure (ESS305, BAY1454032) — Essure is a permanent, minimally invasive, non-hormonal implantable device used for contraception and Adiana sterilization method is a combination of controlled thermal damage to the lining of the fallopian tube followed by insertion of a non-absorbable biocompatible silicone elastomer matrix within the tubal lumen
  Groups: Cohort 1 / Hysteroscopic device placement
Procedure: Tubal ligation — Tubal ligation or tubectomy is a surgical procedure for sterilization in which a woman's fallopian tubes are clamped and blocked, or severed and sealed, either method of which prevents eggs from reaching the uterus for implantation
  Groups: Cohort 2 / Tubal ligation

SUMMARY:
The objective of this study is to describe the proportion of hysterectomy in patients that had undergone sterilization through hysteroscopic device placement and the patients that had undergone sterilization through tubal ligation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 49 years at index date
* Gender: Female
* Diagnosis: Women who underwent hysteroscopic device sterilization procedure
* Diagnosis: Women who underwent tubal ligation sterilization procedure (includes laparoscopic tubal ligation), and salpingectomy

Exclusion Criteria:

* Patients undergoing in-vitro fertilization (IVF) procedures
* Embryo transfer, intrauterine
* Follicle puncture for oocyte retrieval, any method

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 - 49 at index date who underwent hysteroscopic device sterilization procedure or tubal ligation sterilization procedure.
  Index date: Date of sterilization procedure
Sampling Method: Non-Probability Sample
Enrollment: 10578 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients having hysterectomy procedure post-sterilization through hysteroscopic device placement | Retrospective analysis of 10 year period
  The study will also describe sub-outcomes related to post-sterilization hysterectomy procedure including: i. Average time (in days) from index date (sterilization) to hysterectomy ii. Percentage of patients having hysterectomy (abdominal) iii. Percentage of patients having hysterectomy (vaginal) iv. Percentage of patients having hysterectomy (laproscopically assisted vaginal hysterectomy - LAVH) v. Percentage of patients having hysterectomy (abdominal, vaginal and LAVH)
Percentage of patients having hysterectomy procedure post-sterilization through through tubal ligation | Retrospective analysis of 10 year period
  The study will also describe sub-outcomes related to post-sterilization hysterectomy procedure including: i. Average time (in days) from index date (sterilization) to hysterectomy ii. Percentage of patients having hysterectomy (abdominal) iii. Percentage of patients having hysterectomy (vaginal) iv. Percentage of patients having hysterectomy (laproscopically assisted vaginal hysterectomy - LAVH) v. Percentage of patients having hysterectomy (abdominal, vaginal and LAVH)

OTHER OUTCOMES:
Percentage of patients having unintended pregnancy post-sterilization | Retrospective analysis of 10 year period
  Exclusion of any IVF pregnancy, and any pregnancy preceding sterilization
Percentage of patients having unintended ectopic pregnancy post-sterilization | Retrospective analysis of 10 year period
  Exclusion of any IVF pregnancy, and any pregnancy preceding sterilization
Percentage of patients that have salpingectomy (unilateral, bilateral) subsequent to sterilization | Retrospective analysis of 10 year period
Average time in days from sterilization to salpingectomy and Kaplan-Meier-Estimator curve (number of occurrence over time) | Retrospective analysis of 10 year period
Average time in days from sterilization to removal of device inserts other than hysterectomy or salpingectomy and Kaplan-Meier-Estimator curve (number of occurrence over time) | Retrospective analysis of 10 year period
Percentage of patients with repeat sterilization surgery | Retrospective analysis of 10 year period
Average time in days from first sterilization to repeat sterilization surgery and Kaplan-Meier-Estimator curve (number of occurrence over time) | Retrospective analysis of 10 year period
Percentage of patients who undergo a Modified Hysterosalpingogram (HSG) test | Retrospective analysis of 10 year period
Percentage of patients who did not have a Modified HSG and unintentionally got pregnant | Retrospective analysis of 10 year period
Percentage of patients having readmission within 30 days of sterilization | Retrospective analysis of 10 year period
Percentage of patients having removal of device inserts other than hysterectomy or salpingectomy | Retrospective analysis of 10 year period
Percentage of patients who had Modified HSG and got pregnant | Retrospective analysis of 10 year period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- New Jersey, New Jersey, United States